CLINICAL TRIAL: NCT03492112
Title: A Non-randomized Trial to Evaluate a TEst and Treat Intervention Integrating Novel Point-of-care Hepatitis C RNA Testing, Linkage to Nursing Care, and Peer-supported Delivery of HCV Testing and Treatment aMong Current People Who Inject Drugs With HCV Attending Needle and Syringe PrOgrams
Brief Title: A TEst and Treat Intervention aMong Current People Who Inject Drugs With HCV Attending Needle and Syringe PrOgrams
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VHCRP1705
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People attending needle syringe programs in Australia (Experimental): Participants will be screened for Hepatitis C using the Finger-stick whole blood HCV RNA Point of Care GeneXpert. Participants with hepatitis C will be offered treatment with a pan-genotypic DAA HCV therapy- either 12 weeks of sofosbuvir/velpatasvir or 8 weeks of glecaprevir/pibrentasvir.
  Interventions: Device: HCV RNA Point of Care; Drug: Sofosbuvir/velpatasvir; Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Device: HCV RNA Point of Care — Participants attending needle syringe programmes in Australia will be screened for hepatitis C using the finger-stick whole blood GeneXpert HCV RNA cartridge.
  Other Names: GeneXpert System
Drug: Sofosbuvir/velpatasvir — Participants with a detectable HCV RNA will be offered treatment with either glecaprevir/pibrentasvir or sofosbuvir/velpatasvir.
  Other Names: Epclusa
Drug: Glecaprevir/pibrentasvir — Participants with a detectable HCV RNA will be offered treatment with either glecaprevir/pibrentasvir or sofosbuvir/velpatasvir.
  Other Names: Maviret

SUMMARY:
TEMPO is an interventional cohort study recruiting injecting drug users attending needle and syringe programs (NSP) in Australia. Three hundred participants will be invited to on-site HCV testing with NSP integrated care for HCV treatment.

Participants will be screened for HCV using point-of-care testing and HCV positive participants will be offered treatment with Sofosbuvir/Velpatasvir. Of those who initiate treatment, participants will receive weekly peer-based support on-treatment and return at End of Treatment (ETR) and 12 weeks following end of treatment (SVR12) for clinical follow-up.

ELIGIBILITY:
Inclusion criteria

Participants must meet all the following inclusion criteria to be eligible to participate in this study:

1. Participants have voluntarily signed the informed consent form;
2. 18 years of age or older;
3. Current injecting drug use (previous month);
4. HCV RNA positive participants commencing treatment must be eligible to initiate therapy with Sofosbuvir/Velpatasvir; and
5. In the opinion of the Investigator, the participant is suitable for NSP-based HCV treatment delivery.

Exclusion criteria

1) For HCV RNA positive participants commencing treatment:

1. Any clinically significant condition or history known to contraindicate the use of Sofosbuvir/Velpatasvir or would not be suitable for management within a NSP-based treatment setting;
2. Any contraindicated medication in the Sofosbuvir/Velpatasvir product information;
3. Has previous HCV DAA treatment experience
4. Has a fibroscan score > 12.5 Kpa
5. HIV co-infection
6. HBV co-infection
7. Is female and is pregnant or breastfeeding
8. Is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Uptake of HCV DAA therapy among current PWID | 4 Weeks
  Treatment uptake (i.e. proportion of participants initiating DAA therapy)

CONTACTS AND LOCATIONS:
Locations (1):
- NUAA NSP, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grebely J, Gilliver R, McNaughton T, Conway A, Cunningham E, Henderson C, Hadlow B, Molloy K, Doab A, Tillakeratne S, Pepolim L, Harrod ME, Dore GJ, Read P. Single-visit hepatitis C point-of-care testing, linkage to nursing care, and peer-supported treatment among people with recent injecting drug use at a peer-led needle and syringe program: The TEMPO Pilot Study. Int J Drug Policy. 2023 Apr;114:103982. doi: 10.1016/j.drugpo.2023.103982. Epub 2023 Feb 28. PMID 36863287